CLINICAL TRIAL: NCT04437433
Title: A Phase 3, Multicenter, Open-Label 52-Week Extension Study to Evaluate the Long-Term Safety and Tolerability of Oral Atogepant for the Prevention of Migraine in Japanese Participants With Chronic or Episodic Migraine
Brief Title: A Study Evaluating Oral Atogepant for the Prevention of Migraine in Japanese Participants With Chronic or Episodic Migraine
Acronym: JPN ATO OLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3101-306-002
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Results first posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Chronic Migraine; Episodic Migraine
Keywords: Chronic Migraine; Episodic Migraine; Atogepant
MeSH Terms: interventions — atogepant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Atogepant 60 mg Chronic Migraine (Experimental): Participants with chronic migraine (CM) who completed lead-in Study 3101-303-002 (NCT03855137) received atogepant orally as 60 mg tablets once a day (QD) for 52 weeks.
  Interventions: Drug: Atogepant 60 mg
- Atogepant 60 mg Episodic Migraine (Experimental): Participants with episodic migraine (EM) who were newly recruited and met all study entry criteria received atogepant orally as 60 mg tablets once a day (QD) for 52 weeks.
  Interventions: Drug: Atogepant 60 mg

INTERVENTIONS:
Drug: Atogepant 60 mg — Tablets containing 60 mg atogepant

SUMMARY:
This study will evaluate the long-term safety, efficacy and tolerability of atogepant 60 mg daily for the prevention of migraine in Japanese participants with chronic (CM) or episodic migraine (EM).

DETAILED DESCRIPTION:
The study recruited the following 2 cohorts:

3101-303-002 CM Completers: Japanese participants who completed lead-in Study 3101 303-002 (PROGRESS; NCT03855137), a Phase 3, multicenter, randomized, double-blind, placebo controlled, parallel-group study of atogepant for the prevention of CM. All 3101 303-002 CM Completers rolled over at Visit 7 (the end of the double-blind treatment period) of the lead-in study, which functioned as Visit 1 for this study, Study 3101-306-002.

De Novo EM Participants: Japanese participants with EM who were newly recruited for this study at selected sites. Participation began with a 4-week Screening/Baseline period starting at Visit -1, and those who completed the 4-week Screening/Baseline period and met all entry criteria were enrolled into the 52-week open-label treatment period at Visit 1.

ELIGIBILITY:
Inclusion Criteria:

3101-303-002 Completers:

* Eligible participants who completed Visit 7, and Visit 8 if applicable, of the Study 3101-303-002 without significant protocol deviations and who did not experience an adverse event (AE) that, in the investigator's opinion, may indicate an unacceptable safety risk.

De Novo EM Participants:

* Age of the participant at the time of migraine onset < 50 years.
* At least a 1-year history of migraine with or without aura consistent with a diagnosis according to the ICHD-3, 2018.
* History of 4 to 14 migraine days per month on average in the 3 months prior to Visit -1 in the investigator's judgment.
* 4 to 14 migraine days in the 28-day baseline period per eDiary.
* Completed at least 20 out of 28 days in the eDiary during baseline period and is able to read, understand, and complete the study questionnaires and eDiary per investigator's judgment.

Exclusion Criteria:

* Requirement for any medication, diet, or nonpharmacological treatment that is on the list of prohibited concomitant medications or treatments that cannot be discontinued or switched to an allowable alternative medication or treatment.
* Participants with an ECG indicating clinically significant abnormalities at Visit -1 (De Novo EM Participants) or Visit 1 (3103-303-002 Completers).
* Hypertension as defined by sitting systolic BP > 160 mm Hg or sitting diastolic BP > 100 mm Hg at Visit -1 (De Novo EM Participants) or Visit 1 (for all participants)
* Significant risk of self-harm based on clinical interview and responses on the Columbia-Suicide Severity Rating Scale (C-SSRS), or of harm to others in the opinion of the investigator.
* Any clinically significant hematologic, endocrine, cardiovascular, pulmonary, renal, hepatic, gastrointestinal, or neurologic disease.

De Novo EM Participants only:

* Difficulty distinguishing migraine headaches from tension-type or other headaches.
* Has a history of migraine accompanied by diplopia or decreased level of consciousness or retinal migraine as defined by ICHD-3, 2018.
* Has a current diagnosis of chronic migraine, new persistent daily headache, trigeminal autonomic cephalgia (eg, cluster headache), or painful cranial neuropathy as defined by ICHD-3, 2018.
* Has >= 15 headache days per month on average across the 3 months prior to Visit -1 in the investigator's judgment.
* Has >= 15 headache days in the 28-day baseline period per eDiary.
* Usage of opioids or barbiturates > 2 days/month, triptans or ergots >= 10 days/month, or simple analgesics >= 15 days/month in the 3 months prior to Visit -1 per investigator's judgment or during the baseline period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (24):
- Japan (24):
  - Takanoko Hospital /ID# 232723, Matsuyama, Ehime
  - Fukuiken Saiseikai Hospital /ID# 232988, Fukui-shi, Fukui
  - Duplicate_Higashi Sapporo Neurology and Neurosurgery Clinic /ID# 232710, Sapporo, Hokkaido
  - Konan Medical Center /ID# 232922, Kobe, Hyōgo
  - Mito Kyodo General Hospital /ID# 232990, Mito, Ibaraki
  - Atsuchi Neurosurgical Hospital /ID# 232907, Kagoshima, Kagoshima-ken
  - Duplicate_Tokai University Hospital /ID# 233071, Isehara-shi, Kanagawa
  - Fujitsu Clinic /ID# 232717, Kawasaki-shi, Kanagawa
  - Umenotsuji Clinic /ID# 232675, Kochi, Kochi
  - Sendai Headache and Neurology Clinic Medical Corporation /ID# 232677, Sendai, Miyagi
  - Saitama Medical University Hospital /ID# 233017, Iruma-gun, Saitama
  - Saitama Neuropsychiatric Institute /Id# 232711, Saitama-shi, Saitama
  - Japanese Red Cross Shizuoka Hospital /ID# 232992, Shizuoka, Shizuoka
  - Duplicate_Dokkyo Medical University Hospital /ID# 232995, Shimotsuga-gun, Tochigi
  - Niwa Family Clinic /ID# 232713, Chofu-shi, Tokyo
  - Duplicate_Tokyo Headache Clinic /ID# 232715, Shibuya-ku, Tokyo
  - Keio University Hospital /ID# 233030, Shinjuku-ku, Tokyo
  - Duplicate_Nagaseki Headache Clinic /ID# 232719, Kai-shi, Yamanashi
  - DOI Internal Medicine-Neurology Clinic /ID# 232722, Hiroshima
  - Hiroshima Neurology Clinic /ID# 232720, Hiroshima
  - Tanaka Neurosurgical Clinic /ID# 232884, Kagoshima
  - Tatsuoka Neurology Clinic /ID# 232912, Kyoto
  - Tominaga Hospital /ID# 232909, Osaka
  - Shinagawa Strings Clinic /ID# 232908, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=3101-306-002

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of a 52-week open-label treatment period and a 4-week safety follow-up period for all participants.
Period: Overall Study
Arm/Group | Atogepant 60 mg Chronic Migraine | Atogepant 60 mg Episodic Migraine
Started | 155 | 31
Completed | 130 | 28
Not Completed | 25 | 3
Not completed — Met Withdrawal Criteria at Visit 1- Laboratory Values | 7 | 0
Not completed — Met Withdrawal Criteria at Visit 1- ECG | 1 | 0
Not completed — Adverse Event | 9 | 0
Not completed — Lack of Efficacy | 4 | 0
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Protocol Deviation | 0 | 1
Not completed — Other, not specified | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population: all participants who received at least 1 dose of study intervention (atogepant) in this extension study
Groups:
- Total: Total of all reporting groups
Arm/Group | Atogepant 60 mg Chronic Migraine | Atogepant 60 mg Episodic Migraine | Total
Number analyzed (Participants) | 155 | 31 | 186
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (9.47) | 42.4 (11.95) | 43.2 (9.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 29 | 170
  Male | 14 | 2 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 155 | 31 | 186
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 155 | 31 | 186
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least 1 Treatment-Emergent Adverse Event and Treatment-Emergent Serious Adverse Event (TEAEs/TESAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study drug. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent adverse events/treatment-emergent serious adverse events (TEAEs/TESAEs) are defined as any event that began or worsened in severity on or after the first dose of study drug.
Time Frame: From first dose of study drug until 4 weeks following the last dose of study drug (up to 56 weeks)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Atogepant 60 mg Chronic Migraine | Atogepant 60 mg Episodic Migraine
Number analyzed (Participants) | 155 | 31
percentage of participants
  Any TEAE | 88.4 | 90.3
  TESAE | 4.5 | 0.0

2. Secondary Outcome: Percentage of Participants With Potentially Clinically Significant (PCS) Laboratory Values (Chemistry, Hematology, Urinalysis) as Assessed by the Investigator
Description: Clinical laboratory test values are considered PCS if they meet either the lower-limit or higher-limit PCS criteria defined in the categories below. The percentage of participants with PCS laboratory values are summarized for hematology, chemistry, and urinalysis.
Time Frame: From first dose of study drug until 4 weeks following the last dose of study drug (up to 56 weeks)
Population: Safety population: all participants who received at least 1 dose of study intervention (atogepant) in this extension study. Number analyzed are participants with data available for analyses of the specific category.
Measure: Number; unit: percentage of participants
Arm/Group | Atogepant 60 mg Chronic Migraine | Atogepant 60 mg Episodic Migraine
Number analyzed (Participants) | 155 | 31
percentage of participants
  Basophils (10^9/L): > 2.0 x Upper Limit of Normal (ULN) | 0.0 | 0.0
  Eosinophils (10^9/L): > 2.0 x Upper Limit of Normal (ULN) | 0.0 | 0.0
  Erythrocytes, Hematology (10^12/L): < 0.9 x Lower Limit of Normal (LLN) | 3.2 | 3.2
  Erythrocytes, Hematology (10^12/L): > 1.1 x Upper Limit of Normal (ULN) | 0.0 | 0.0
  Hematocrit (RATIO): < 0.9 x Lower Limit of Normal (LLN): number analyzed (Participants) | 152 | 31
  Hematocrit (RATIO): < 0.9 x Lower Limit of Normal (LLN) | 0.0 | 0.0
  Hematocrit (RATIO): > 1.1 x Upper Limit of Normal (ULN): number analyzed (Participants) | 152 | 31
  Hematocrit (RATIO): > 1.1 x Upper Limit of Normal (ULN) | 0.0 | 0.0
  Hemoglobin (g/L): < 0.9 x Lower Limit of Normal (LLN): number analyzed (Participants) | 150 | 31
  Hemoglobin (g/L): < 0.9 x Lower Limit of Normal (LLN) | 3.3 | 0.0
  Hemoglobin (g/L): > 1.1 x Upper Limit of Normal (ULN): number analyzed (Participants) | 150 | 31
  Hemoglobin (g/L): > 1.1 x Upper Limit of Normal (ULN) | 0.0 | 0.0
  Leukocytes, Hematology (10^9/L): < 0.9 x Lower Limit of Normal (LLN): number analyzed (Participants) | 148 | 29
  Leukocytes, Hematology (10^9/L): < 0.9 x Lower Limit of Normal (LLN) | 12.8 | 17.2
  Leukocytes, Hematology (10^9/L): > 1.5 x Upper Limit of Normal (ULN): number analyzed (Participants) | 148 | 29
  Leukocytes, Hematology (10^9/L): > 1.5 x Upper Limit of Normal (ULN) | 0.0 | 0.0
  Lymphocytes (10^9/L): < 0.7 x Lower Limit of Normal (LLN) | 1.9 | 0.0
  Lymphocytes (10^9/L): > 1.3 x Upper Limit of Normal (ULN) | 0.0 | 0.0
  Monocytes (10^9/L): < 0.5 x Lower Limit of Normal (LLN) | 0.0 | 0.0
  Monocytes (10^9/L): > 2.0 x Upper Limit of Normal (ULN) | 0.0 | 0.0
  Neutrophils (10^9/L): < 0.7 x Lower Limit of Normal (LLN): number analyzed (Participants) | 153 | 31
  Neutrophils (10^9/L): < 0.7 x Lower Limit of Normal (LLN) | 2.6 | 3.2
  Neutrophils (10^9/L): > 1.3 x Upper Limit of Normal (ULN): number analyzed (Participants) | 153 | 31
  Neutrophils (10^9/L): > 1.3 x Upper Limit of Normal (ULN) | 0.7 | 0.0
  Platelets (10^9/L): < 0.5 x Lower Limit of Normal (LLN) | 0.0 | 0.0
  Platelets (10^9/L): > 1.5 x Upper Limit of Normal (ULN) | 1.3 | 0.0
  Alanine Aminotransferase (U/L): ≥ 3.0 x Upper Limit of Normal (ULN) | 5.8 | 0.0
  Albumin (g/L): < 0.8 x Lower Limit of Normal (LLN) | 0.0 | 0.0
  Albumin (g/L): > 1.2 x Upper Limit of Normal (ULN) | 0.0 | 0.0
  Alkaline Phosphatase (U/L): ≥ 3.0 x Upper Limit of Normal (ULN) | 0.6 | 0.0
  Aspartate Aminotransferase (U/L): ≥ 3.0 x Upper Limit of Normal (ULN) | 3.2 | 0.0
  Bicarbonate (mmol/L): < 0.9 x Lower Limit of Normal (LLN) | 0.6 | 3.2
  Bicarbonate (mmol/L): > 1.1 x Upper Limit of Normal (ULN) | 0.0 | 0.0
  Bilirubin, Chemistry (umol/L): ≥ 1.5 x Upper Limit of Normal (ULN) | 0.6 | 0.0
  Calcium (mmol/L): < 0.9 x Lower Limit of Normal (LLN) | 0.0 | 0.0
  Calcium (mmol/L): > 1.1 x Upper Limit of Normal (ULN) | 0.0 | 0.0
  Chloride (mmol/L): < 0.9 x Lower Limit of Normal (LLN) | 0.0 | 0.0
  Chloride (mmol/L): > 1.1 x Upper Limit of Normal (ULN) | 0.0 | 0.0
  Cholesterol (mmol/L): > 1.6 x Upper Limit of Normal (ULN) | 0.0 | 0.0
  Creatine Kinase (U/L): > 2.0 x Upper Limit of Normal (ULN) | 2.6 | 0.0
  Creatinine (umol/L): > 1.5 x Upper Limit of Normal (ULN) | 0.0 | 0.0
  Glomerular Filtration Rate, Estimated (mL/min/1.73): < 60 mL/min/1.73m^2: number analyzed (Participants) | 154 | 30
  Glomerular Filtration Rate, Estimated (mL/min/1.73): < 60 mL/min/1.73m^2 | 1.9 | 3.3
  Glucose, Chemistry (mmol/L): < 0.8 x Lower Limit of Normal (LLN) | 1.9 | 0.0
  Glucose, Chemistry (mmol/L): > 2.0 x Upper Limit of Normal (ULN) | 0.0 | 0.0
  Lactate Dehydrogenase (U/L): > 3.0 x Upper Limit of Normal (ULN) | 0.6 | 0.0
  Phosphate (mmol/L): < 0.9 x Lower Limit of Normal (LLN) | 0.0 | 0.0
  Phosphate (mmol/L): > 1.1 x Upper Limit of Normal (ULN) | 0.0 | 0.0
  Potassium (mmol/L): < 0.9 x Lower Limit of Normal (LLN) | 0.0 | 0.0
  Potassium (mmol/L): > 1.1 x Upper Limit of Normal (ULN) | 0.0 | 0.0
  Protein, Chemistry (g/L): < 0.9 x Lower Limit of Normal (LLN) | 0.0 | 0.0
  Protein, Chemistry (g/L): > 1.1 x Upper Limit of Normal (ULN) | 0.0 | 0.0
  Sodium (mmol/L): < 0.9 x Lower Limit of Normal (LLN) | 0.0 | 0.0
  Sodium (mmol/L): > 1.1 x Upper Limit of Normal (ULN) | 0.0 | 0.0
  Urate (umol/L): > 1.2 x Upper Limit of Normal (ULN) | 0.0 | 0.0
  Urea Nitrogen (mmol/L): > 1.5 x Upper Limit of Normal (ULN) | 0.0 | 0.0
  Glucose, Urinalysis: At least 1+: number analyzed (Participants) | 152 | 30
  Glucose, Urinalysis: At least 1+ | 1.3 | 0.0
  Protein, Urinalysis: At least 1+: number analyzed (Participants) | 143 | 30
  Protein, Urinalysis: At least 1+ | 28.7 | 26.7
  Specific Gravity: > 1.1 x Upper Limit of Normal (ULN) | 0.0 | 0.0
  pH: < 0.9 x Lower Limit of Normal (LLN) | 0.0 | 0.0
  pH: > 1.1 x Upper Limit of Normal (ULN) | 0.0 | 0.0

3. Secondary Outcome: Percentage of Participants With Potentially Clinically Significant (PCS) Electrocardiograms (ECGs) Findings as Assessed by the Investigator
Description: 12-lead ECGs were performed at select study visits.
Time Frame: Week -4 (De Novo Participants), Day 1 (3101-303-002 Completers Only), Weeks 12, 24, 36, and 52
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Atogepant 60 mg Chronic Migraine | Atogepant 60 mg Episodic Migraine
Number analyzed (Participants) | 155 | 31
percentage of participants
  PR Interval (msec): ≥ 250 | 0.0 | 0.0
  QRS Duration (msec): ≥ 150 | 0.0 | 0.0
  QTcF Interval (msec): > 500 | 0.0 | 0.0
  QTcF Interval (msec): Increase from Baseline of > 60 | 0.0 | 0.0

4. Secondary Outcome: Percentage of Participants With Potentially Clinically Significant (PCS) Vital Sign Measurements as Assessed by the Investigator
Description: Potentially Clinically Significant post-Baseline vital sign values are summarized for categories: systolic and diastolic blood pressures [sitting and standing], pulse rate [sitting and standing], and weight.
Time Frame: From first dose of study drug until 4 weeks following the last dose of study drug (up to 56 weeks)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Atogepant 60 mg Chronic Migraine | Atogepant 60 mg Episodic Migraine
Number analyzed (Participants) | 155 | 31
percentage of participants
  Sitting, Standing Systolic Blood Pressure (mmHg): ≥ 180 and increase from Baseline of ≥ 20 | 0.0 | 0.0
  Sitting, Standing Systolic Blood Pressure (mmHg): ≤ 90 and decrease from Baseline of ≥ 20 | 5.8 | 9.7
  Sitting, Standing Diastolic Blood Pressure (mmHg): ≥ 105 and increase from Baseline of ≥ 15 | 4.5 | 3.2
  Sitting, Standing Diastolic Blood Pressure (mmHg): ≤ 50 and decrease from Baseline of ≥ 15 | 0.6 | 0.0
  Sitting, Standing Pulse Rate (bpm): ≥ 120 and increase from Baseline of ≥ 15 | 0.6 | 0.0
  Sitting, Standing Pulse Rate (bpm): ≤ 50 and decrease from baseline of ≥ 15 | 1.3 | 0.0
  Weight (kg): Increase from Baseline of ≥ 7% | 4.5 | 3.2
  Weight (kg): Decrease from Baseline of ≥ 7% | 32.9 | 25.8
  Orthostatic Systolic Blood Pressure (mmHg): ≤ -20: number analyzed (Participants) | 153 | 31
  Orthostatic Systolic Blood Pressure (mmHg): ≤ -20 | 12.4 | 6.5
  Orthostatic Diastolic Blood Pressure (mmHg): ≤ -15 | 3.9 | 0.0
  Orthostatic Pulse Rate (bpm): ≥ 25 | 4.5 | 6.5

5. Secondary Outcome: Percentage of Participants With Most Severe Suicidal Ideation and Suicidal Behavior as Assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) During the Open-Label Treatment Period
Description: The C-SSRS is a clinician-rated instrument that reports the severity of both suicidal ideation and behavior. Suicidal ideation is classified on a 5-item scale: 1 (wish to be dead), 2 (nonspecific active suicidal thoughts), 3 (active suicidal ideation with any methods [not plan] without intent to act), 4 (active suicidal ideation with some intent to act, without specific plan), and 5 (active suicidal ideation with specific plan and intent). Suicidal behavior is classified on a 5-item scale: 0 (no suicidal behavior), 1 (preparatory acts or behavior), 2 (aborted attempt), 3 (interrupted attempt), and 4 (actual attempt). More than 1 classification can be selected provided they represent separate episodes. (Minimum total score 0, maximum total score 5; higher total scores indicate more suicidal ideation and/or suicidal behavior).
Time Frame: From first dose of study drug until the last dose of study drug (up to 52 weeks)
Population: Safety population: all participants who received at least 1 dose of study intervention (atogepant) in this extension study.; participants with available data
Measure: Number; unit: percentage of participants
Arm/Group | Atogepant 60 mg Chronic Migraine | Atogepant 60 mg Episodic Migraine
Number analyzed (Participants) | 155 | 31
percentage of participants
  No suicidal ideation | 98.1 | 100
  Suicidal ideation | 1.3 | 0.0
  Most severe suicidal ideation: Active suicidal ideation with specific plan and intent | 0.0 | 0.0
  Most severe suicidal ideation: Active suicidal ideation with some intent to act, w/out specific plan | 0.0 | 0.0
  Most severe suicidal ideation: Active suicidal ideation w/ any method (not plan) w/out intent to act | 0.0 | 0.0
  Most severe suicidal ideation: Non-specific active suicidal thoughts | 0.6 | 0.0
  Most severe suicidal ideation: Wish to be dead | 0.6 | 0.0
  No suicidal behavior: number analyzed (Participants) | 154 | 31
  No suicidal behavior | 100 | 100.0
  Suicidal behavior: number analyzed (Participants) | 154 | 31
  Suicidal behavior | 0.0 | 0.0
  Most severe suicidal behavior: Actual attempt: number analyzed (Participants) | 154 | 31
  Most severe suicidal behavior: Actual attempt | 0.0 | 0.0
  Most severe suicidal behavior: Interrupted attempt: number analyzed (Participants) | 154 | 31
  Most severe suicidal behavior: Interrupted attempt | 0.0 | 0.0
  Most severe suicidal behavior: Aborted attempt: number analyzed (Participants) | 154 | 31
  Most severe suicidal behavior: Aborted attempt | 0.0 | 0.0
  Most severe suicidal behavior: Preparatory acts or behavior: number analyzed (Participants) | 154 | 31
  Most severe suicidal behavior: Preparatory acts or behavior | 0.0 | 0.0
  Completed Suicide | 0.0 | 0.0
  Non-suicidal self-injurious behavior | 0.0 | 0.0

6. Secondary Outcome: Percentage of Participants With Most Severe Suicidal Ideation and Suicidal Behavior as Assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) During the Safety Follow-Up Period
Description: as for outcome 5
Time Frame: Up to 4 weeks following the last dose of study drug
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Atogepant 60 mg Chronic Migraine | Atogepant 60 mg Episodic Migraine
Number analyzed (Participants) | 155 | 31
percentage of participants
  No suicidal ideation: number analyzed (Participants) | 154 | 31
  No suicidal ideation | 100 | 93.5
  Suicidal ideation: number analyzed (Participants) | 154 | 31
  Suicidal ideation | 0.0 | 0.0
  Most severe suicidal ideation: Active suicidal ideation with specific plan and intent: number analyzed (Participants) | 154 | 31
  Most severe suicidal ideation: Active suicidal ideation with specific plan and intent | 0.0 | 0.0
  Most severe suicidal ideation: Active suicidal ideation with some intent to act, w/out specific plan: number analyzed (Participants) | 154 | 31
  Most severe suicidal ideation: Active suicidal ideation with some intent to act, w/out specific plan | 0.0 | 0.0
  Most severe suicidal ideation: Active suicidal ideation w/ any method (not plan) w/out intent to act: number analyzed (Participants) | 154 | 31
  Most severe suicidal ideation: Active suicidal ideation w/ any method (not plan) w/out intent to act | 0.0 | 0.0
  Most severe suicidal ideation: Non-specific active suicidal thoughts: number analyzed (Participants) | 154 | 31
  Most severe suicidal ideation: Non-specific active suicidal thoughts | 0.0 | 0.0
  Most severe suicidal ideation: Wish to be dead: number analyzed (Participants) | 154 | 31
  Most severe suicidal ideation: Wish to be dead | 0.0 | 0.0
  No suicidal behavior: number analyzed (Participants) | 154 | 31
  No suicidal behavior | 100 | 93.5
  Suicidal behavior: number analyzed (Participants) | 154 | 31
  Suicidal behavior | 0.0 | 0.0
  Most severe suicidal behavior: Actual attempt: number analyzed (Participants) | 154 | 31
  Most severe suicidal behavior: Actual attempt | 0.0 | 0.0
  Most severe suicidal behavior: Interrupted attempt: number analyzed (Participants) | 154 | 31
  Most severe suicidal behavior: Interrupted attempt | 0.0 | 0.0
  Most severe suicidal behavior: Aborted attempt: number analyzed (Participants) | 154 | 31
  Most severe suicidal behavior: Aborted attempt | 0.0 | 0.0
  Most severe suicidal behavior: Preparatory acts or behavior: number analyzed (Participants) | 154 | 31
  Most severe suicidal behavior: Preparatory acts or behavior | 0.0 | 0.0
  Completed Suicide | 0.0 | 0.0
  Non-suicidal self-injurious behavior | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from the time informed consent was signed to the end of the study. The median time on follow-up was 392 days for the Atogepant 60 mg Chronic Migraine group, 421 days for the Atogepant 60 mg Episodic Migraine group, and 392 days for all participants.
Groups:
- Total: Participants received atogepant orally as 60 mg tablets once a day (QD) for 52 weeks.
Arm/Group | Atogepant 60 mg Chronic Migraine | Atogepant 60 mg Episodic Migraine | Total
All-Cause Mortality (participants affected / at risk) | 0/155 | 0/31 | 0/186
Serious Adverse Events (participants affected / at risk) | 7/155 | 0/31 | 7/186
Other Adverse Events (participants affected / at risk) | 108/155 | 24/31 | 132/186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atogepant 60 mg Chronic Migraine (N=155) | Atogepant 60 mg Episodic Migraine (N=31) | Total (N=186)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
APPENDICITIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 1 (1)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
MIGRAINE (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atogepant 60 mg Chronic Migraine (N=155) | Atogepant 60 mg Episodic Migraine (N=31) | Total (N=186)
DRY EYE (Eye disorders) | 4 (4) | 2 (2) | 6 (6)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 6 (7) | 2 (3) | 8 (10)
CONSTIPATION (Gastrointestinal disorders) | 17 (17) | 4 (5) | 21 (22)
DIARRHOEA (Gastrointestinal disorders) | 8 (9) | 2 (2) | 10 (11)
STOMATITIS (Gastrointestinal disorders) | 3 (6) | 2 (2) | 5 (8)
MALAISE (General disorders) | 9 (11) | 1 (1) | 10 (12)
PYREXIA (General disorders) | 52 (68) | 2 (2) | 54 (70)
COVID-19 (Infections and infestations) | 1 (1) | 6 (7) | 7 (8)
CYSTITIS (Infections and infestations) | 11 (12) | 1 (1) | 12 (13)
GINGIVITIS (Infections and infestations) | 1 (1) | 2 (2) | 3 (3)
NASOPHARYNGITIS (Infections and infestations) | 18 (19) | 12 (19) | 30 (38)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 10 (14) | 3 (3) | 13 (17)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 7 (10) | 2 (2) | 9 (12)
DECREASED APPETITE (Metabolism and nutrition disorders) | 5 (5) | 2 (2) | 7 (7)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 8 (8) | 2 (2) | 10 (10)
MYALGIA (Musculoskeletal and connective tissue disorders) | 10 (14) | 0 (0) | 10 (14)
HEADACHE (Nervous system disorders) | 8 (11) | 1 (1) | 9 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/33/NCT04437433/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-26): https://cdn.clinicaltrials.gov/large-docs/33/NCT04437433/SAP_001.pdf